CLINICAL TRIAL: NCT00290745
Title: Primary Hormonal Therapy for Ductal Carcinoma in Situ: Exploration of a Novel Approach to the Clinical Management of Noninvasive Breast Cancer
Brief Title: Tamoxifen or Letrozole in Treating Women With Ductal Carcinoma in Situ
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 017513; UCSF-H10367-19435-05 (Other: University of California, San Francisco); NCI-2011-01273 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); CDR0000465205 (Other: University of California, San Francisco)
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Results first posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
Keywords: breast cancer in situ; ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Carcinoma, Intraductal, Noninfiltrating | interventions — Letrozole; Tamoxifen; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- tamoxifen or letrozole (Experimental): tamoxifen or letrozole work in treating women with ductal carcinoma in situ
  Interventions: Drug: letrozole; Drug: tamoxifen citrate; Procedure: conventional surgery; Procedure: neoadjuvant therapy

INTERVENTIONS:
Drug: letrozole
Drug: tamoxifen citrate
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using tamoxifen or letrozole may fight breast cancer by blocking the use of estrogen by the tumor cells or by lowering the amount of estrogen the body makes.

PURPOSE: This clinical trial is studying how well tamoxifen or letrozole work in treating women with ductal carcinoma in situ.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical response in women with estrogen receptor-positive ductal carcinoma in situ (DCIS) treated with neoadjuvant hormonal therapy comprising tamoxifen or letrozole, by evaluating the maximal change in tumor diameter on mammography and MRI following treatment.
* Identify those cellular antigens which are altered by hormonal therapy.
* Determine which cellular antigens are predictive of clinical response to hormonal therapy.
* Evaluate whether genomic changes or gene expression in DCIS are altered by hormonal therapy and find candidate genes which are correlated with response to treatment.

OUTLINE: This is a pilot study.

Patients who are premenopausal receive oral tamoxifen once daily for 3 months in the absence of unacceptable toxicity. Patients who are post menopausal receive oral letrozole once daily for 3 months in the absence of unacceptable toxicity.

After 3 months of hormonal therapy, patients undergo lumpectomy or mastectomy.

After completion of study treatment, patients are followed every 6 months for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of ductal carcinoma in situ (DCIS) on core biopsy
* No evidence of contralateral breast disease or palpable masses on breast examination
* No presence or suspicion of invasive cancer, including contralateral invasive cancer, on core biopsy and MRI
* No documented ipsilateral axillary adenopathy
* Planning to undergo lumpectomy or mastectomy
* Estrogen receptor (ER)-positive tumor by immunohistochemistry

PATIENT CHARACTERISTICS:

* Female patient
* Premenopausal or postmenopausal

  * Postmenopausal is defined by any of the following:

    * No spontaneous menses for >= 1 year
    * Bilateral oophorectomy
    * Radiation castration and amenorrheic for >= 3 months
    * Follicle-stimulating hormone (FSH) > 20 IU/L AND off all hormonal therapy (e.g., hormone replacement therapy or birth control pills) for >= 1 month
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No co-morbidities contraindicating the use of tamoxifen, including any of the following:

  * Prior history of thrombotic events
  * History of hypercoagulable state
  * History of endometrial hyperplasia
  * Abnormal vaginal bleeding
* No history of contrast dye-related allergies/reactions
* No history of metal-containing prostheses or implants

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2002-02-19 (Actual); Primary Completion 2009-07-31 (Actual); Study Completion 2011-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Shelley Hwang, MD, MPH, Principal Investigator — University of California, San Francisco; Frederic M. Waldman, MD, PhD, Principal Investigator — University of California, San Francisco; Nola M. Hylton, PhD, Principal Investigator — University of California, San Francisco; Rita Mukhtar, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen YY, DeVries S, Anderson J, Lessing J, Swain R, Chin K, Shim V, Esserman LJ, Waldman FM, Hwang ES. Pathologic and biologic response to preoperative endocrine therapy in patients with ER-positive ductal carcinoma in situ. BMC Cancer. 2009 Aug 18;9:285. doi: 10.1186/1471-2407-9-285. PMID 19689789
- [Background] Swain RS, Chen YY, Wa C, et al.: Pathologic and biologic response to neoadjuvant anti-estrogen (AE) therapy in patients with ductal carcinoma in situ (DCIS). [Abstract] United States and Canadian Academy of Pathology 95th Annual Meeting, February 11-17, 2006, Atlanta, GA. A-186, 2006.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients seeking treatment at the University of California, San Francisco (UCSF) Breast Care Center and Kaiser Permanente for a diagnosis of DCIS were approached by their physicians at their discretion, and if fitting the eligibility criteria were asked to participate in the study.
Groups:
- Tamoxifen or Letrozole: tamoxifen or letrozole work in treating women with ductal carcinoma in situ
  letrozole
  tamoxifen citrate
  conventional surgery
  neoadjuvant therapy
Period: Overall Study
Arm/Group | Tamoxifen or Letrozole
Started | 79
Completed | 67
Not Completed | 12
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 2
Not completed — Surgery after 3 months for progression | 3
Not completed — Baseline MRI not available | 3

BASELINE CHARACTERISTICS:
Population: Baseline data collected for evaluable patients only
Arm/Group | Tamoxifen or Letrozole
Number analyzed (Participants) | 67
Age, Continuous [Median (Full Range); unit: years] | 62.9 [49.7 to 83.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 54
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 67
Nuclear Grade [Count of Participants; unit: Participants] — The nuclear grade describes how closely the nuclei of cancer cells look like the nuclei of normal breast cells. In general, the higher the nuclear grade, the more abnormal the nuclei are and the more aggressive the tumor cells tend to be. The nuclear grade is also a part of overall tumor grade.
  Participants
    Low (Grade 1) | 8
    Intermediate (Grade 2) | 31
    High (Grade 3) | 27
    Indeterminate | 1
Hormone receptor status [Count of Participants; unit: Participants] — Hormone receptors are proteins, found in and on breast cells, that pick up hormone signals telling the cells to grow. A cancer is called estrogen-receptor-positive (ER+) if it has receptors for estrogen. This suggests that cancer cells may receive signals from estrogen that could promote their growth. The cancer is progesterone-receptor-positive (PgR+) if it has progesterone receptors. This means that cancer cells may receive signals from progesterone that could promote their growth. If the cancer is hormone-receptor-negative (ER- or PgR-) then no receptors are present,
  Participants
    ER+ / PgR+ | 55
    ER+/(PgR- or PgR Unknown) | 10
    ER-/PgR+ | 2

OUTCOME MEASURES:

1. Primary Outcome: Median Change in 6-month Tumor Volume Compared to Baseline Using Mammography
Description: Change in size of Ductal Carcinoma in situ (DCIS) for participants on hormonal therapy, as determined by mammography are determined by (1) largest diameter of tumor, as visualized on mammography (2) extent of disease on mammography (3) quantification of mammographically-detected change from baseline to 6-month and used to generate the change in tumor volume of mammographic extent of disease from baseline. Since values were not normally distributed, the median change was calculated, and Wilcoxon sign rank tests were used to evaluate the significance of these changes
Time Frame: Baseline and 6 months
Population: Only 54 patients had evaluable mammograms at 6 months
Measure: Median (Inter-Quartile Range); unit: change in tumor volume (mm)
Arm/Group | Tamoxifen or Letrozole
Number analyzed (Participants) | 54
change in tumor volume (mm) | -5.0 [-10.4 to 0.4]
Statistical Analysis 1: Comparison: Tamoxifen or Letrozole; Change in Tumor volume between baseline and Month 6; Test type: Other; p = 0.07, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Median Change in 6-month Tumor Volume Compared to Baseline Using Magnetic Resonance Imaging (MRI)
Description: Change in size of Ductal Carcinoma in situ (DCIS) on hormonal therapy, as determined by MRI are determined by (1) largest diameter of tumor, as visualized on MRI (2) extent of disease on MRI (3) quantification of MR-detected change from baseline to 6-month and used to generate the change in tumor volume of MRI extent of disease from baseline. Since values were not normally distributed, the median change was calculated, and Wilcoxon sign rank tests were used to evaluate the significance of these changes.
Time Frame: Baseline and 6 months
Measure: Median (Inter-Quartile Range); unit: change in tumor volume (cm3)
Arm/Group | Tamoxifen or Letrozole
Number analyzed (Participants) | 67
change in tumor volume (cm3) | -0.8 [-1.95 to 0.35]
Statistical Analysis 1: Comparison: Tamoxifen or Letrozole; Change in Tumor volume between baseline and Month 6; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Responders to Neoadjuvant Therapy at Month 3
Description: MRI volume response at each time point was classified as follows: 90% image-complete response (ICR90) is defined as a >90% reduction in tumor volume, 80% image-complete response (ICR80) is defined as an 81-90% reduction in tumor volume , partial response (PR) is defined as a 20-80% reduction in tumor volume, and sustained disease or progressive disease (SD/PD) defined as a <20% reduction or increase in volume.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tamoxifen or Letrozole
Number analyzed (Participants) | 67
Participants
  ICR90 | 13
  ICR80 | 10
  PR | 27
  SD/PD | 17

4. Secondary Outcome: Number of Responders to Neoadjuvant Therapy at Month 6
Description: as for outcome 3
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tamoxifen or Letrozole
Number analyzed (Participants) | 67
Participants
  ICR90 | 22
  ICR80 | 7
  PR | 26
  SD/PD | 12

5. Secondary Outcome: Median Reduction in Tumor Volume by Estrogen Receptor Hormone (ER H-) Quartile Group
Description: Tumor volume changes between baseline and surgery were calculated at month 6 and compared across baseline ER Hormone (H-) Score quartile. The ER H- scores are a percentage that tells you how many cells out of 100 stain positive for hormone receptors. Each participant is assigned an ER H- score at baseline with the full score range between 0 (none have receptors) and 100 (all have receptors). The participants were grouped into quartiles (four equal groups) based on their baseline ER H- score. ER H- score and the reduction in tumor volume from baseline to month 6 was measured for each quartile group.
Time Frame: Baseline and 6 months
Population: Only 46 participants had both evaluable ER scores at baseline and evaluable month 6 scans
Measure: Median (Inter-Quartile Range); unit: decrease in tumor volume (cm^3)
Arm/Group | Tamoxifen or Letrozole
Number analyzed (Participants) | 46
decrease in tumor volume (cm^3)
  Baseline ER Score quartile = 0-25: number analyzed (Participants) | 12
  Baseline ER Score quartile = 0-25 | -58.8 [-141.6 to 24]
  Baseline ER Score quartile = 26-50: number analyzed (Participants) | 11
  Baseline ER Score quartile = 26-50 | -70.3 [-91.2 to 49.4]
  Baseline ER Score quartile = 51-75: number analyzed (Participants) | 12
  Baseline ER Score quartile = 51-75 | -80.3 [-92.1 to -68.5]
  Baseline ER Score quartile = 76-100: number analyzed (Participants) | 11
  Baseline ER Score quartile = 76-100 | -71.1 [-85.75 to -56.45]
Statistical Analysis 1: Comparison: Tamoxifen or Letrozole; Test type: Other; p = 0.538, Kruskal-Wallis

6. Secondary Outcome: Median Reduction in Tumor Volume by PgR H-score by Quartile Group
Description: Tumor volume changes between baseline and surgery were calculated at month 6 and compared across baseline PgR Hormone (H-) Score quartile. The PgR H-scores are a percentage that tells you how many cells out of 100 stain positive for hormone receptors. Each participant is assigned a PgR H- score at baseline with the full PgR H score ranges between 0 (none have receptors) and 100 (all have receptors). The participants were grouped into quartiles (four equal groups) based on their baseline PgR H- score and the reduction in tumor volume from baseline to month 6 was measured for each quartile group.
  A wilcoxon sign rank tests were used to evaluate the significance of these changes
Time Frame: Baseline and 6 months
Population: Only 45 participants had both evaluable PgR scores at baseline and evaluable month 6 scans
Measure: Median (Inter-Quartile Range); unit: reduction in tumor volume (cm^3)
Arm/Group | Tamoxifen or Letrozole
Number analyzed (Participants) | 45
reduction in tumor volume (cm^3)
  Baseline PgR Score Quartile = 0-25: number analyzed (Participants) | 12
  Baseline PgR Score Quartile = 0-25 | -69.1 [-103.7 to -34.5]
  Baseline PgR Score Quartile = 26-50: number analyzed (Participants) | 11
  Baseline PgR Score Quartile = 26-50 | -45.8 [-130.95 to 39.95]
  Baseline PgR Score Quartile = 51-75: number analyzed (Participants) | 13
  Baseline PgR Score Quartile = 51-75 | -69.6 [-85.65 to -56.65]
  Baseline PgR Score Quartile = 76-100: number analyzed (Participants) | 9
  Baseline PgR Score Quartile = 76-100 | -96.2 [-106.2 to -86.2]
Statistical Analysis 1: Comparison: Tamoxifen or Letrozole; Test type: Other; p = 0.02, Kruskal-Wallis

7. Secondary Outcome: Median Reduction in Tumor Volume by Ki-67 Average Score
Description: Tumor volume changes between baseline and surgery were calculated at month 6 by Baseline Ki-67 Average Score which is divided into 2 groups: (1) <=10% or (2) >10% to 100%. In est results, the Ki-67 findings expressed as a percentage with less than 10% considered low Ki-67 expression and > than 10% or higher considered high. A "high" score means that the breast tumor is more likely to be aggressive and spread quickly. A wilcoxon sign rank tests were used to evaluate the significance of these changes
Time Frame: Baseline and 6 months
Population: Only 45 participants had both evaluable Ki-67 scores at baseline and evaluable month 6 scan
Measure: Median (Inter-Quartile Range); unit: reduction in tumor volume (cm^3)
Arm/Group | Tamoxifen or Letrozole
Number analyzed (Participants) | 45
reduction in tumor volume (cm^3)
  Baseline Ki67 Average <=10%: number analyzed (Participants) | 22
  Baseline Ki67 Average <=10% | -73.0 [-98.45 to -47.55]
  Baseline Ki67 Average > 10%: number analyzed (Participants) | 25
  Baseline Ki67 Average > 10% | -70.3 [-88.55 to -52.05]
Statistical Analysis 1: Comparison: Tamoxifen or Letrozole; Test type: Other; p = 0.714, Kruskal-Wallis

8. Secondary Outcome: Correlation Between Pathologic Tumor Size at Radiographic (MRI) Tumor Size
Description: Correlations between pathologic tumor size and maximum diameters of baseline and 6-month MRI extent of disease were evaluated using Spearman correlation coefficient measure of association. The Spearman's rank-order correlation (rs) measures the strength and direction of association between two variables. The Spearman correlation coefficient, rs, can take values from +1 to -1 where a value of +1 indicates a perfect association, an rs of 0 indicates no association and an rs of -1 indicates a perfect negative association. The closer rs is to 0, the weaker the association.
Time Frame: 6 months
Measure: Number; unit: Spearman correlation coefficient (rs)
Arm/Group | Tamoxifen or Letrozole
Number analyzed (Participants) | 67
Spearman correlation coefficient (rs) | 0.46
Statistical Analysis 1: Comparison: Tamoxifen or Letrozole; Test type: Other; p = 0.001, Kruskal-Wallis

9. Secondary Outcome: Correlation Between Pathologic Tumor Size and Mammographic Tumor Size
Description: Correlations between pathologic tumor size and maximum diameters of baseline and pre-surgical mammographic extent of disease were evaluated using Spearman correlation coefficient measure of association. The Spearman's rank-order correlation (rs) measures the strength and direction of association between two variables. The Spearman correlation coefficient, rs, can take values from +1 to -1 where a value of +1 indicates a perfect association, an rs of 0 indicates no association and an rs of -1 indicates a perfect negative association. The closer rs is to 0, the weaker the association.
Time Frame: 6 months
Population: Only 54 patients had evaluable mammograms at 6 months
Measure: Number; unit: Spearman correlation coefficient (rs)
Arm/Group | Tamoxifen or Letrozole
Number analyzed (Participants) | 54
Spearman correlation coefficient (rs) | 0.02
Statistical Analysis 1: Comparison: Tamoxifen or Letrozole; Test type: Other; p = 0.906, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: All good cause efforts to retrieve the serious adverse event and non-serious adverse event data have been exhausted. Adverse event data are no longer accessible per institutional and contractual guidelines for record retention and hence not available to be reported.
Arm/Group | Tamoxifen or Letrozole
All-Cause Mortality (participants affected / at risk) | 0/67
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
All good cause efforts to retrieve the serious adverse event and non-serious adverse event data have been exhausted. Adverse event data are no longer accessible per institutional and contractual guidelines and hence not available to be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No